CLINICAL TRIAL: NCT00933595
Title: Longitudinal Studies of HIV-Associated Lung Infections and Complications (Lung HIV)
Acronym: LHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Johns Hopkins University (Other); Johns Hopkins Bloomberg School of Public Health (Other); New York University (Other); Ohio State University (Other); University of California, San Francisco (Other); University of Colorado, Denver (Other); University of Pittsburgh (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 652; 3R01HL090331-05S1 (NIH)
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Complications; HIV Infections
Keywords: HIV; Lung
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Smoking Cessation (Experimental): The overall smoking cessation rate for the intervention is 18.8 at 3 months, 13.1 at 6 months and 10.0 at 12 months.
  Interventions: Other: Smoking Cessation

INTERVENTIONS:
Other: Smoking Cessation — A Motivational Interview session (~40-50 minutes) will be delivered by a trained nurse coordinator.
  Treatment with varenicline (1 mg daily during week 1 (pre-quit week) followed by 1 mg twice daily for weeks 2-12)or nicotine replacement therapy (21 mg of a skin patch + nicotine gum 4 mg ad lib added for breakthrough craving up to 20 pieces/day.

SUMMARY:
The Lung HIV goal is to facilitate the data and specimen collection efforts of eight individual HIV and pulmonary studies that operate under the direction of the NHLBI. The Lung HIV study will build on existing studies to facilitate the start-up of new projects to further the understanding of the relationship between pulmonary disease and HIV infection. There is only one clinical trial being performed in this network at Ohio State University and it will be reported here.

DETAILED DESCRIPTION:
The Ohio State University Clinical Research Center (CRC), Patient Selection

Study Intervention Subjects:

365 HIV+ male and female smokers will be enrolled to the study and will be recruited over a two - four year period.

Inclusion criteria

1. 18 years of age and older
2. Diagnosis of HIV (Since the vast majority of our subjects will be recruited through the OSU Infectious disease clinics and HIV clinical research unit documentation of HIV status will not be a problem)
3. Self-reported smoking (≥ 5 cigarettes per day to avoid inclusion of occasional, 'social' users and 'chippers');
4. Able and willing to provide informed written consent.

Exclusion criteria:

1. Inability to provide informed consent
2. Inability to understand spoken English
3. Currently diagnosed interstitial lung disease (i.e. sarcoidosis, idiopathic pulmonary fibrosis) or lung cancer.

Control Subjects Group A:

We will utilize normal subjects for the control study for the Diffusion Capacity of Lung for Carbon Monoxide (DLCO) and Diffusion capacity of Lung for Nitric Oxide (DLNO), recruited from the general population. We will recruit 5 males and 5 females in each decade of life from 21-30, 31-40, 41-50, 51-60, 61-70 (TOTAL= 50 subjects).

Inclusion criteria

1. 21-70 years of age and older
2. HIV Seronegative
3. Able and willing to provide informed written consent.

Exclusion criteria:

1. Inability to provide informed consent
2. Inability to understand spoken English
3. Current smoker or have smoked in the last 10 years or have a > 10 pack year history of smoking.
4. Currently diagnosed interstitial lung disease (i.e. sarcoidosis, idiopathic pulmonary fibrosis) or lung cancer.

Control Subjects Group B:

We will utilize normal subjects for the control study for DLCO and DLNO, recruited from the general population. We will recruit 5 males and 5 females in each decade of life from 21-30, 31-40, 41-50, 51-60, 61-70 (TOTAL= 50 subjects).

Inclusion criteria

1. 21-70 years of age and older
2. HIV Seronegative
3. Current or former smoker with at least a 5 pack year history of smoking
4. Able and willing to provide informed written consent.

Exclusion criteria:

1. Inability to provide informed consent
2. Inability to understand spoken English
3. Currently diagnosed interstitial lung disease (i.e. sarcoidosis, idiopathic pulmonary fibrosis) or lung cancer.

ELIGIBILITY:
Inclusion Criteria

Men and women at the AIDS Clinical Trials Unit(ACTU) will be eligible to participate if they meet four criteria: (a) 18 years of age and older; and (b) diagnosis of HIV; and (c) self-reported smoking on a daily basis; and (d) provide informed written consent.

Exclusion criteria

Persons who meet one or more of the following criteria will be excluded from the study: (a) persons with active psychosis or impaired mental status as judged by the clinic staff and confirmed with a Mini-Mental Status Exam); (b) unable to understand spoken English; (c) age less than 18 years.

Rationale: Persons with cognitive impairment may participate in the study if they are able to provide consent and answer questionnaire questions. No reason is identified to exclude persons with this characteristic. No special risks are posed to cognitively impaired persons who are able to provide consent. Persons who have active psychoses or impaired mental status as judged by the clinic staff and confirmed with a Mini-Mental Status Exam are not able to provide informed written consent and are unlikely to benefit from the treatment. These persons will be referred to appropriate mental health services and invited to participate when their mental status has improved.

Persons who are unable to understand spoken English would not be able to complete the assessments or benefit from the treatments. Less than 1% of the clinic population will be excluded on this basis. However, persons excluded from the study on this basis will be referred for standard smoking cessation treatment delivered in their native tongue. These community resources may be identified through the Ohio State University Nursing Center for Tobacco Intervention.

Younger adolescents (<18 years) will not be invited to participate in the study because we believe that they require treatments that are qualitatively different from those designed for older adolescents and adults. The treatments that will be evaluated in the proposed research are well suited to older adolescents and adults, but not developmentally tailored to younger adolescents. Less than 1% of the clinic population will be excluded on this basis. Most HIV+ children living in Columbus, Ohio receive HIV medical care through the F.A.C.E.S. outpatient clinic at Columbus Children's Hospital. Standard, age appropriate, smoking cessation treatment is available through the Health and Wellness Center at Columbus Children's Hospital. In the unlikely circumstance that a child <18 years of age wishes to participate in the proposed study, s/he will be referred to Health and Wellness Center at Children's Hospital for treatment or the Ohio State University Nursing Center for Tobacco Intervention for age appropriate smoking cessation community resources.

Pregnant women may not be included as subjects. While smoking during pregnancy is an important modifiable cause of poor pregnancy outcomes, little information is available on the safety or efficacy of varenicline. Therefore, participants who are pregnant will be excluded as subjects. Also, women who are breast-feeding will be excluded.

Other persons who are unable to use varenicline will be allowed to participate in the study but will not receive the varenicline component of treatment. A history and physical examination will be conducted as a component of the baseline evaluation.

People that have kidney problems or undergo kidney dialysis will not take the study drug, but will be given the option to take nicotine replacement therapy.

All persons excluded from the study will have the opportunity to receive smoking cessation treatment. We will provide referrals for treatment as clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To develop and evaluate a specialized smoking cessation intervention for the treatment of nicotine dependence in HIV-seropositive smokers. | 5 years

SECONDARY OUTCOMES:
To examine the effects of smoking cessation on the course of lung function decline, the prevalence of respiratory symptoms and the occurrence/progression of emphysema in a cohort of HIV-seropositive individuals. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Peavy, MD, Study Director — NHLBI Project Officer
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Crothers K, Thompson BW, Burkhardt K, Morris A, Flores SC, Diaz PT, Chaisson RE, Kirk GD, Rom WN, Huang L; Lung HIV Study. HIV-associated lung infections and complications in the era of combination antiretroviral therapy. Proc Am Thorac Soc. 2011 Jun;8(3):275-81. doi: 10.1513/pats.201009-059WR. PMID 21653528
- Available data/document: Individual Participant Data Set: LUNG-HIV — http://biolincc.nhlbi.nih.gov/studies/lung_hiv/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/lung_hiv/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/lung_hiv/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/lung_hiv/